CLINICAL TRIAL: NCT02780440
Title: Home Mirror Therapy: A Randomized Control Study Comparing Unimanual and Bimanual Mirror Therapy for Improved Hand Function Post-stroke
Brief Title: Comparing Unimanual and Bimanual Mirror Therapy for Upper Limb Recovery Post Stroke
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 14-01859
Record Dates: First submitted 2016-05-19; First posted 2016-05-23 (Estimated); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Cerebral Vascular Accident (CVA); Stroke
Keywords: Post Stroke Recovery; Mirror Therapy; Unimanual mirror therapy; Bimanual mirror therapy; Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control Group: Subjects will participate in standard occupational therapy rehabilitation protocol plus a traditional home based exercise program.
  Interventions: Behavioral: Traditional Home Based Exercise Program
- Experimental Group 1: Subjects will participate in standard rehabilitation protocol plus unimanual home based mirror therapy program
  Interventions: Behavioral: Unimanual Home Based Mirror Therapy Program
- Experimental Group 2: Subjects will participate in standard rehabilitation protocol plus bimanual home based mirror therapy program.
  Interventions: Behavioral: Bimanual Home Based Mirror Therapy Program

INTERVENTIONS:
Behavioral: Traditional Home Based Exercise Program — Subjects in the control group will receive a traditional home Occupational Training exercise program as per conventional OT guidelines with the same home program duration.
  Groups: Control Group
Behavioral: Unimanual Home Based Mirror Therapy Program — The affected hand will remain still in the mirror box, the unaffected hand will perform the exercises while the subject watches the mirror reflection.
  Groups: Experimental Group 1
Behavioral: Bimanual Home Based Mirror Therapy Program — The affected hand in the mirror box will best mimic the unaffected hand, while also watching the mirror reflection.
  Groups: Experimental Group 2

SUMMARY:
The purpose of this randomized controlled study is to

1. Examine the feasibility of a home Mirror therapy (MT) program in the NYC metropolitan area;
2. Evaluate the effectiveness of home MT versus traditional home exercise program; and
3. Evaluate the superiority of unimanual or bimanual MT intervention protocols for chronic stroke subjects with moderate hand deficits. Subjects from occupational therapy at the Ambulatory Care Center of NYU Langone Center with a diagnosis of cerebral vascular accident (CVA) or stroke will be divided into three (3) groups:

   * Control Group subjects will participate in standard occupational therapy rehabilitation protocol plus a traditional home based exercise program.
   * Experimental group 1 subjects will participate in standard rehabilitation protocol plus unimanual home based mirror therapy program
   * Experimental group 2 subjects will participate in standard rehabilitation protocol plus bimanual home based mirror therapy program.

ELIGIBILITY:
Inclusion Criteria:

* First time unilateral stroke > 3 months post stroke.
* Cognitively be able to follow direction
* Cognitively be able to consent to participation in research study
* Moderate/severe deficits as per the Fugl-Meyer assessment score from 10-50 and the ability to grasp and release a small towel or washcloth.

Exclusion Criteria:

* Complex medical problems, that would render the subject unable to participate in an extensive home program
* History of pre-existing neurological or psychiatric diseases, orthopedic conditions of the upper limbs, or peripheral nerve injuries that render the subject unable to sit or to move either upper limb
* Hearing and vision impairments which may impede subjects participation in the home program
* Perceptual deficits such as apraxia, neglect, or agnosias as per clinical evaluation which may impede subjects participation in the home program
* Botox injection in affected arm/hand within 3 months
* Global aphasia that may interfere with understanding instruction for testing or home exercise program.

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants included in the study will be those referred to outpatient occupational therapy at the Ambulatory Care Center of NYU Langone Center with a diagnosis of cerebral vascular accident (CVA) or stroke.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2014-11; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment (FMA) | Baseline to Six (6) Weeks
  Gold Standard to evaluate and measure recovery in patients with hemiplegia post stroke.
Grip strength | Baseline to Six (6) Weeks
  Grip strength is important to measure as it is correlated with stroke recovery.
Action Research Arm Test (ARAT) | Baseline to Six (6) Weeks
  An interview based tool that measures a subject's perceived difficulty with the use of their arm/hands with activities of daily living post-stroke.
Stroke Impact Scale Version 3.0 | Baseline to Six (6) Weeks
  A subjective standardized 59-items 8 domain questionnaire assessing health status post-stroke.

CONTACTS AND LOCATIONS:
Overall Officials: Steve Vanlew, MD, Principal Investigator — New York University Medical School
Locations (1):
- New York University School of Medicine, New York, New York, United States

REFERENCES:
- [Derived] Geller D, Nilsen DM, Quinn L, Van Lew S, Bayona C, Gillen G. Home mirror therapy: a randomized controlled pilot study comparing unimanual and bimanual mirror therapy for improved arm and hand function post-stroke. Disabil Rehabil. 2022 Nov;44(22):6766-6774. doi: 10.1080/09638288.2021.1973121. Epub 2021 Sep 19. PMID 34538193